CLINICAL TRIAL: NCT04480489
Title: The Efficacy of Immersive 360-degree Video in Improving Spatial Orientation Among Medical Students
Brief Title: Testing Efficacy of VR in Medical Education
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-5565
Record Dates: First submitted 2020-07-17; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Virtual Reality and Medical Education

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial. Pre-clerkship (year 1 and 2) medical students from the University of Toronto Faculty of Medicine will be recruited to take part in the study. Participants will complete a baseline questionnaire collecting data quantifying key potentially confounding factors such as previous 360 videos, previous visits to Toronto Western Hospital, physical gait disability, and navigation experience.
  A 2x2 study design will be used to implement counterbalancing as a way to control for two important sources of systematic variation in this type of study: practice and boredom effects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): In Group A, students will first perform Task 1 (walk from anesthesia lounge to the day surgery unit) using intervention 1 (using the virtual reality video) first, then Task 2 (walk from anesthesia lounge to the pre-operative clinic) using intervention 2 (using the traditional 2D video).
  Interventions: Other: VR; Other: Traditional
- group B (Active Comparator): In Group B, students will first perform Task 1 (follow route 1: walk from anesthesia lounge to the day surgery unit) using intervention 2 (using the traditional 2D video) first, then Task 2 (follow route 2: walk from anesthesia lounge to the pre-operative clinic) using intervention 1 (using the virtual reality video).
  Interventions: Other: VR; Other: Traditional

INTERVENTIONS:
Other: VR — Task 1: Students will be first taken to the anesthesia lounge. Here the students will receive VR instructions on how to navigate Route 1 (i.e. they will watch a 360-degree immersive video using Samsung VR headset).
  Task 2: After completing the Route 1 walkthrough, the same group will be given traditional instructions (2D video) on navigating Route 2, followed by an observed walkthrough of Route 2.
  Students in the arm "Group A" will perform Task 1 using VR and then Task 2 using Traditional video. Meanwhile students in the arm "Group B" will perform Task 1 using Traditional video and Task 2 using VR
Other: Traditional — Task 1: Students will be first taken to the anesthesia lounge. Here the students will receive traditional instructions (2D video) on how to navigate Route 1.
  Task 2: After completing the Route 1 walkthrough, the same group will be given VR instructions on how to navigate Route 2, followed by an observed walkthrough of Route 2.
  Students in the arm "Group A" will perform Task 1 using VR and then Task 2 using Traditional video. Meanwhile students in the arm "Group B" will perform Task 1 using Traditional video and Task 2 using VR

SUMMARY:
Recent emergence and commercialization of immersive virtual reality (VR) shows great promise in its application to medical education. While the technology is rapidly developing, we don't yet know how we learn in an immersive environment. As a result, this study will investigate how medical students at the University of Toronto learn from immersive 360-degree video (i.e. VR) when compared to standard 2D video. The task to learn will be hospital (i.e. Toronto Western Hospital) navigation.

DETAILED DESCRIPTION:
The recent emergence and commercialization of immersive virtual reality (VR) shows great promise in its application to medical education. While several surgical, critical care, and procedural 'virtual reality simulators' are described, very few immersive VR experiences that use 360-degree videos have been described (Alakar et al., 2016; Zhu et al., 2014). 360-degree video is a form of virtual reality that shows video content in a globe creating a sense of immersion and realism that is not possible in standard 2D-videos. The videos are viewed using a virtual reality headset capable of displaying the 360-degree content. Among the few studies that do describe immersive learning experiences in medical training, very few have explored the modality from a pedagogical perspective (Barsom et al., 2017; Cha et al, 2006). It is still unclear whether learning via an immersive experience through 360-degree videos is better than traditional methods such as 2D videos.

The use of traditional 2D video is quite well established in medical education as it enhances knowledge transfer, communication skills, attitude formation, and appeals to learners with various learning styles (Abraham et al, 2011; de Leng et al., 2007). Videos are commonly used for clinical skills training as they provide standardized and consistent learning experiences (Flores et al., 2010; Knowles et al., 2001). They can also be used as resources for 'just-in-time' learning, where students preview content by watching videos before attending didactic or hands-on sessions. Patient case videos allow for rare clinical scenarios to be available to students in perpetuity (Gagliano, 1988). The use of video has allowed for the delivery of educational content in both asynchronous and synchronous (i.e. live or real-time) formats allowing for streaming of video to distant locations with real-time dialogue at all sites (Bridge et al., 2009; Gandsas et al., 2004). These advantages of video have enabled the rapid expansion of some medical schools to multiple hospitals. As medical students rotate through these sites during their clinical years, they often face the challenge of adjusting to unfamiliar environments. Anecdotal as well as survey feedback from our site suggests that unfamiliarity with a new environment induces anxiety among trainees and may result in some 'false' starts on the first day of the rotations. Furthermore, the unfamiliarity may cause students to get lost and arrive late to their clinical assignments. Current solutions include text-based directions for way-finding and orientation, which are at times are supplemented by photographs and standard 2-dimensional video. The realism of 360-degree videos may provide a sense of direction with better wayfinding skills because it will allow the learner to explore and 'experience' the depicted location. To date, there is no study reported comparing 2D with 360-degree video on wayfinding and the orientation experience for medical students.

The use of video to assist with wayfinding and orientation exists but is not currently reported in the literature. Spofford et al. (2012) conducted a randomized controlled trial to evaluate the utility of standard lecture and 2D video in orienting students to the anesthesia machine and the operating room setup. The orientation 2D video group performed significantly better with higher post-test scores but scored lower on satisfaction as students preferred the traditional lecture. The study did not assess the utility of orientation videos for wayfinding. Furthermore, the efficacy in improving spatial orientation, reducing anxiety, or enhancing the orientation process is not well known.

Hypothesis: 360-degree videos will enhance spatial orientation of medical students by:

1. Improving way-finding and sense of orientation
2. Conferring a sense of presence
3. Increasing level of satisfaction with the learning experience
4. Decreasing anxiety with a new environment

Methods:

This will be a prospective randomized controlled trial. Pre-clerkship (year 1 and 2) medical students from the University of Toronto Faculty of Medicine will be recruited to take part in the study. Participants will complete a baseline questionnaire collecting data quantifying key potentially confounding factors such as previous 360 videos, previous visits to Toronto Western Hospital, physical gait disability, and navigation experience.

Students will be randomized to two groups (see below) and given video orientation for each route. It takes approximately 4 minutes to walk each one.

Route 1: Conference room 2nd floor to the Day Surgery Unit on the 4th floor. Route 2: Anesthesia lounge on 2nd floor to preoperative assessment clinic on the ground floor to the operating rooms on the 2nd floor

The goal of having each group complete different routes is to assess internal validity within each group when given traditional vs. VR instructions. Group 1 and 2 will also be compared to assess which learning method is superior.

ELIGIBILITY:
Inclusion Criteria:

* Pre-clerkship (year 1 and 2) medical students from the University of Toronto Faculty of Medicine.

Exclusion Criteria:

* Any medical students who have had experience visiting Toronto Western Hospital for personal reasons or previous coursework, shadowing, research, or clinical rotations.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-28 (Estimated); Primary Completion 2020-10-02 (Estimated); Study Completion 2020-10-23 (Estimated)

PRIMARY OUTCOMES:
Time assessment | End of the study (2 hours)
  A research assistant will follow and time how long it takes the medical student to travel from the starting to end point.

SECONDARY OUTCOMES:
Distance assessment | End of the study (2 hours)
  The number of steps and distance travelled will be measured using a standardized pedometer.
Number of wrong turns/wrong floors/doors entered | End of the study (2 hours)
  Way finding corrective measures
Number of times student asks for help. | End of the study (2 hours)
  Way finding corrective measures

OTHER OUTCOMES:
Student measure of satisfaction | End of the study (2 hours)
  In addition to objective assessments, we will have a subjective questionnaire that participants will complete at the end of the study to indicate their comfort with spatial orientation and level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: AHTSHAM NIAZI, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to preserve student privacy and confidentiality throughout the course of the study and the feedback they share at the end of the study. The students however will be provided access to both the VR and the traditional 2D hospital orientation videos once the study is complete.